CLINICAL TRIAL: NCT02996773
Title: A Phase I/Ib Study of Haploidentical Bone Marrow Transplant With Post-Transplant Cyclophosphamide and/or Bendamustine
Brief Title: Haploidentical BMT With Post-Transplant Cyclophosphamide and Bendamustine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1609876907
Record Dates: First submitted 2016-12-01; First posted 2016-12-19 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia; Lymphoma,Non-Hodgkin; Lymphoma, Hodgkin; Lymphoma, Follicular; Marginal Zone Lymphoma; Large Cell Lymphoma; Mantle-Cell Lymphoma; Gray Zone Lymphoma; Burkitt Lymphoma; High Risk Undifferentiated Acute Leukemia
Keywords: high-risk malignancies; Lymphoma; Haploidentical; Bone Marrow Transplant (BMT); Post-transplant; myeloablative (MAC); reduced intensity conditioning (RIC); haploidentical hematopoietic cell transplantation (HHCT); Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma; Mycobacterium avium-intracellulare Infection; Leukemia | interventions — Bendamustine Hydrochloride; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide and Bendamustine (Experimental): Experimental: Cyclophosphamide and Bendamustine Control: Cyclophosphamide
  Interventions:
  * Drug: Bendamustine
  * Drug: Cyclophosphamide
  Interventions: Drug: Bendamustine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Bendamustine — After transplant, given intravenously on day +4 as part of Phase Ib.
  Other Names: BEN
Drug: Cyclophosphamide — After transplant, given intravenously on day +3 as part of Phase 1b.
  Other Names: CY

SUMMARY:
The purpose of this study is to evaluate the safety of progressively substituting day +3 and +4 post-transplant cyclophosphamide (PT-CY) with post-transplant bendamustine (PT-BEN) in myeloablative (MAC) haploidentical hematopoietic cell transplantation (HHCT) for patients with hematological malignancies.

The goal of the Phase 1 component of the study is to evaluate the safety of progressively substituting post-transplant cyclophosphamide (PT-CY) given on Days +3 and +4 with bendamustine (PT-BEN). The Phase I component of the study has been completed.

The Phase Ib component of the study will continue to evaluate the safety and efficacy of subjects who receive PT-BEN on Days +3 and +4 at the maximum tolerated dose determined by Phase I. The Phase Ib component of the study has been completed.

Approximately, 18-36 subjects will be treated as part of Phase I and 15 as part of Phase Ib. Approximately 18 subjects will be used as controls, subjects that receive no PET-BEN, for direct comparison. Total, approximately 38-56 treatment and control patients and 38-56 donor subjects will be enrolled.

DETAILED DESCRIPTION:
This study will follow the standard-of-care bone marrow transplant (BMT), with the only exception being to progressively substitute post-transplant cyclophosphamide (on Days +3 and +4 after BMT) with bendamustine. Six dose levels were planned for the Phase I component of the study, consisting of a combination of sequentially reduced doses of cyclophosphamide (PT-CY) and increased doses of bendamustine (PT-BEN) initially on Day +4 after BMT, followed by the same sequential reduction and increase on Day +3. An interim analysis was performed after cohort 3 was completed in Phase I and included a preliminary comparison between treatment and control groups. Phase Ib will evaluate patients treated with PT-CY on day +3 and PT-BEN on day +4.

Control patients will be patients that have declined to participate in the main trial but will receive haploidentical BMT with the current standard of two days of PT-CY (and no PT-BEN) and will be consented for the immune monitoring studies only.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written consent/assent for the trial.
* Diagnosed with one of the following high-risk malignancies, which require hematopoietic cell transplantation (HCT) but do not have an available Human Leukocyte Antigen (HLA)-matched related or unrelated donor or acceptable cord blood
* High risk acute lymphoblastic leukemia (ALL) in 1st complete remission (CR1) or greater
* High risk acute myelogenous leukemia (AML) in CR1 or greater
* High risk undifferentiated acute leukemia
* High risk myelodysplastic syndrome (MDS)
* Chronic Myelogenous Leukemia (CML) failing or intolerant to Tyrosine Kinase Inhibitors (TKIs) or in accelerated, blastic phase, or in second or subsequent chronic phase
* Lymphoma, (Hodgkin and Non-Hodgkins Lymphoma including marginal zone, follicular lymphoma, chemotherapy-sensitive large-cell, mantle cell lymphoma, gray zone, and Burkitt's lymphoma in remission).
* At least one haploidentical related donor is available for bone marrow harvest.
* Molecular based HLA typing for the HLA-A, -B, -Cw, beta chain (-DRB1) and - DQ Beta 1 Locus (DQB1loci) to the resolution is needed to establish haploidentity.
* A minimum match of 5/10 is required.
* No availability of an 8/8 HLA-matched related or unrelated donor or clinical urgency for transplant (e.g., needed within 4-8 weeks) at which time an acceptable unrelated donor will not be available.

Exclusion Criteria:

* Refractory acute leukemia (>5% blasts) or progressive disease
* Untreated or progressive central nervous system leukemia
* Refractory to chemotherapy lymphoma
* Co-morbidities precluding patient's ability to tolerate BMT
* Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) > 5 x upper limit of normal (ULN)
* Bilirubin > 2 x ULN
* Creatinine greater than >2 x ULN for age or creatinine clearance/glomerular filtration rate (GFR) <40 ml/min/1.73m2
* Pulmonary function: Diffusing capacity of the lung for carbon monoxide (DLCO) < 40% of normal or O2 Sat <92%
* Cardiac: left ventricular ejection fraction <35%
* Active infection at time of hospital admission of Haplo BMT
* Documented fungal infection or highly suspected and receiving treatment for presumed fungal infection within 3 months of BMT
* HIV positive
* Karnofsky score (adults) < 60% or Lansky score < 50% (pediatrics).
* Positive pregnancy test for girls post menarche or women of childbearing age.
* Severe psychiatric illness or mental deficiency making compliance to treatment unlikely and/or informed consent impossible.
* Any reason, at the investigator's discretion, that the participation of the patient in this protocol would not be in patient's best interest, or where the patient would be unable to adhere to the study requirements.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Safety in regards to engraftment, incidence and grade of acute and chronic graft-versus-host-disease, graft failure, infections, relapse, and non-relapse mortality post-haploidentical bone marrow transplantation. | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups
  Examine the effects of PT-BEN on immune reconstitution following human haploidentical BMT.

SECONDARY OUTCOMES:
Incidence of regimen-related organ toxicities | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Incidence of acute GvHD | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Severity of acute GvHD | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Incidence of chronic GvHD | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Extent of chronic GvHD | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Incidence of graft failure | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Infection risk | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
  Immune reconstitution will be studied prospectively. Viral and fungal prophylaxis and treatment will be done according to our BMT programs guidelines
Infection severity | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
  Immune reconstitution will be studied prospectively. Viral and fungal prophylaxis and treatment will be done according to our BMT programs guidelines
Overall patient survival | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
Immune reconstitution following haploidentical BMT | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
  T cell immune reconstitution (CD4, cluster of differentiation 8 (CD8), Treg, NK), B cell and myeloid cell reconstitution will be evaluated serially until 6 months post-BMT
Incidence of bacterial, fungal and viral infections/reactivations | Change from baseline to 3 years. Interim analysis will be performed after cohort 3 and cohort 6 in Phase 1, and include preliminary evaluation of treatment and control groups]
  Gather data on Incidence of bacterial, fungal and viral infections/reactivations

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Katsanis, MD, Principal Investigator — The University of Arizona Cancer Center
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Result] Baker FL, Stokes J, Cracchiolo MJ, Davini D, Simpson RJ, Katsanis E. Impact of post-transplant cyclophosphamide with bendamustine on immune reconstitution in young patients undergoing T-cell replete haploidentical bone marrow transplantation: results from a phase Ia/Ib clinical trial. Front Immunol. 2025 Apr 9;16:1568862. doi: 10.3389/fimmu.2025.1568862. eCollection 2025. PMID 40270968
- [Result] Katsanis E, Stea B, Kovacs K, Truscott L, Husnain M, Khurana S, Roe DJ, Simpson RJ. Feasibility and Efficacy of Partially Replacing Post-Transplantation Cyclophosphamide with Bendamustine in Pediatric and Young Adult Patients Undergoing Haploidentical Bone Marrow Transplantation. Transplant Cell Ther. 2022 Jul;28(7):390.e1-390.e10. doi: 10.1016/j.jtct.2022.04.015. Epub 2022 Apr 20. PMID 35460929
- [Result] Katsanis E, Sapp LN, Reid SC, Reddivalla N, Stea B. T-Cell Replete Myeloablative Haploidentical Bone Marrow Transplantation Is an Effective Option for Pediatric and Young Adult Patients With High-Risk Hematologic Malignancies. Front Pediatr. 2020 Jun 9;8:282. doi: 10.3389/fped.2020.00282. eCollection 2020. PMID 32582591
- [Result] Katsanis E, Maher K, Roe DJ, Simpson RJ. Progressive substitution of posttransplant cyclophosphamide with bendamustine: A phase I study in haploidentical bone marrow transplantation. EJHaem. 2020 May 26;1(1):286-292. doi: 10.1002/jha2.20. eCollection 2020 Jul. PMID 35847727
- [Result] Katsanis E, Sapp LN, Varner N, Koza S, Stea B, Zeng Y. Haploidentical Bone Marrow Transplantation with Post-Transplant Cyclophosphamide/Bendamustine in Pediatric and Young Adult Patients with Hematologic Malignancies. Biol Blood Marrow Transplant. 2018 Oct;24(10):2034-2039. doi: 10.1016/j.bbmt.2018.06.007. Epub 2018 Jun 14. PMID 29908231